CLINICAL TRIAL: NCT02321709
Title: A Randomized, Double-blind, Placebo-controlled Study Of Safety, Tolerability, And Pharmacokinetics Of Repeated Ascending Subcutaneous Doses Of SAR113244 And Pharmacodynamics Of Single Dose Of SAR113244 In Male And Female Lupus Patients
Brief Title: Multiple Ascending Dose Study To Assess The Safety Profile Of SAR113244 Versus Placebo In Lupus Male And Female Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: TDR11407; 2014-001690-13 (EudraCT Number); U1111-1154-6184 (Other: UTN)
Record Dates: First submitted 2014-12-05; First posted 2014-12-22 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-04

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- SAR113244 cohort 1 (Experimental): Two administrations of dosage 1 SAR113244 or placebo subcutaneous dose (Q4 weeks)
  Interventions: Drug: SAR113244; Drug: placebo
- SAR113244 cohort 2 (Experimental): Two administrations of dosage 2 SAR113244 or placebo subcutaneous dose (Q4 weeks)
  Interventions: Drug: SAR113244; Drug: placebo
- SAR113244 cohort 3 (Experimental): Two administrations of dosage 3 SAR113244 or placebo subcutaneous dose (Q4 weeks)
  Interventions: Drug: SAR113244; Drug: placebo

INTERVENTIONS:
Drug: SAR113244 — Pharmaceutical form:solution for injection Route of administration: subcutaneous
Drug: placebo — Pharmaceutical form:solution for injection Route of administration: subcutaneous

SUMMARY:
Primary Objective:

To assess the tolerability and safety of SAR113244 in male and female lupus patients after every 4 (Q4) weeks repeated ascending subcutaneous doses of SAR113244.

Secondary Objectives:

To assess in male and female lupus patients:

* The pharmacokinetics of SAR113244.
* The pharmacodynamics of SAR113244 for the following disease-related parameters:

  * Safety of Estrogens in Lupus Erythematosus National Assessment - Systemic Lupus Erythematosus Disease Activity Index (SELENA-SLEDAI) score, British Isles Lupus Assessment Group (BILAG) score (if applicable), BILAG-Based Composite Lupus Assessment (BICLA) (if applicable), systemic lupus erythematosus responder index (SRI) (if applicable), Lupus-quality of life (QoL) and Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue, anti-double stranded deoxyribonucleic acid antibody (anti-dsDNA Ab) and anti-nuclear antibody levels (ANA) and plasma complement levels (C3, C4), erythrocyte sedimentation (SED) rate and C-reactive protein.
  * Peripheral blood B and T cells subsets.

DETAILED DESCRIPTION:
The total duration of screening to end of study per subject is 20 weeks with post-study observation on Day 226 for anti-drug antibody assessment (for patients with positive anti-drug antibody at end of study only).

ELIGIBILITY:
Inclusion criteria:

* Male or female patients, between 18 and 75 years of age, inclusive.
* Clinical diagnosis of systemic lupus erythematosus (SLE) by American College Rheumatology criteria.
* Autoantibody-posititve.
* On active and stable SLE disease.

Exclusion criteria:

* Pregnant and nursing.
* Have received treatment with investigational drugs in the 4 months prior to the screening or 5 half-lives of the drug, whichever is longer.
* Have received intravenous or oral cyclophosphamide within 180 days of Day 0. Severe active lupus nephritis or chronic renal insufficiency.
* Active or chronic, severe neuropsychiatric lupus.
* Acute, recent (within 4 weeks of screening), chronic or frequently recurring infection(s), except minor infection.
* Have current drug or alcohol abuse or dependence.
* Have a historically positive test or test postitive at screening for HIV, hepatitis B, or hepatitis C.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-11; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events and treatment-emergent adverse events | Up to 16 weeks after inclusion
Change in physical examination, body weight, vital signs and laboratory parameters | Up to 16 weeks after inclusion
Safety and tolerability (erythema, swelling, degree of itching, and present pain intensity at injection site by measuring diameter and qualitative assessment) | Up to 16 weeks after inclusion

SECONDARY OUTCOMES:
Assessment of pharmacokinetic parameter - maximum concentration (Cmax) | Up to D113 after inclusion
Assessment of pharmacokinetic parameter - time of maximum concentration (Tmax) | Up to D113 after inclusion
Assessment of pharmacokinetic parameter - area under curve 0-4 weeks (AUC0-4w) | Up to D113 after inclusion
Assessment of pharmacokinetic parameter - time of the last point with quantifiable concentration (tlast) and terminal elimination half-life (t1/2z) | Up to D113 after inclusion
Assessment of pharmacokinetic parameter - lowest concentration of drug before the next dose (Ctrough) | Up to D113 after inclusion
Assessment of pharmacokinetic parameter - apparent total body clearance (CLss/F) | Up to D113 after inclusion
Assessment of pharmacokinetic parameter - absorption-dependent apparent volume of distribution at steady state (Vss/F) | Up to D113 after inclusion
Number of participants with anti-SAR113244 antibody titers | Up to D226 after inclusion
Pharmacodynamic parameter changes | Up to D113 after inclusion
Pharmacodynamic parameters: peripheral blood B and T cells subsets | Up to D85 after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number 276001, Berlin, Germany